CLINICAL TRIAL: NCT06475235
Title: A Pilot Study of Pembrolizumab in Combination With Chemotherapy in Newly Diagnosed Primary Central Nervous System Lymphoma
Brief Title: Pembrolizumab + Chemotherapy in Newly Diagnosed PCNSL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lakshmi Nayak, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-246
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Primary Central Nervous System Lymphoma
Keywords: Lymphoma; Primary Central Nervous System Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab; Immunoglobulin G; Methotrexate; Temozolomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Induction Treatment: (Experimental): Participants will be enrolled and will complete procedures as follows, starting at Dose Level 0 for Methotrexate and Temozolomide:
  * Baseline visit with assessments and imaging.
  * Imaging on cycles 3 and 6 only.
    * Cycles 1 through 3:
      ---Days 3 and 10 of 14 day cycle: Predetermined dose of Rituximab 1x daily.
    * Cycles 1, 3, 5, and 7:
      ---Days 7 through 11 of 14 day cycle: Predetermined dose of Temozolomide 1x daily.
    * Cycles 1 through 8:
      ---Day 1 of 14 day cycle: Predetermined dose of Methotrexate 1x daily.
    * Cycles 1, 4, 7
    * Day 10 of 14 day cycle: Predetermined dose of Pembrolizumab 1x daily. Treatment will de-escalate per protocol if greater than or equal to 2 out of 6 participants experience a dose-limiting toxicity.
  Interventions: Drug: Pembrolizumab; Drug: Methotrexate; Drug: Temozolomide; Drug: Rituximab
- Consolidation Treatment: (Experimental): 4-8 weeks after the completion of Induction Cycle 8, the study doctor will determine if it is appropriate to move on to consolidation therapy and participants will complete:
  * Imaging every other cycle.
  * Cycles 1 through 15:
    * Day 1 of 42 day cycle: Lumbar puncture
    * Day 1 of 42 day cycle: Predetermined dose of Pembrolizumab 1x daily.
  * End of treatment visit with lumbar puncture and imaging.
  * Follow up
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Humanized immunoglobin G4 monoclonal antibody, 4 mL vials, via intravenous infusion (into the vein) per protocol.
  Other Names: Keytruda; MK-3475; Humanized X PD-1 mAb (H409A11) IgG4
Drug: Methotrexate — Anti-metabolite, 50 mL vials, via intravenous infusion per protocol.
  Other Names: MTX
  Arms: Induction Treatment:
Drug: Temozolomide — Alkylating agent, 5, 20, 100, 140, 180, or 250 mg capsules, taken orally per protocol.
  Other Names: Temodar; Temodal
  Arms: Induction Treatment:
Drug: Rituximab — Anti-CD20 antibody, 10 or 50 mL single-use vials, via intravenous infusion per standard of care.
  Other Names: Riabni; Rituxan; Ruxience; Truxima
  Arms: Induction Treatment:

SUMMARY:
This research study is studying if the investigational drug, Pembrolizumab, in combination with chemotherapy helps primary central nervous system lymphoma with acceptable side effects.

This research study involves a combination of the below drugs:

* Pembrolizumab (a type of monoclonal antibody)
* Methotrexate (a type of anti-metabolite)
* Temozolomide (a type of alkylating agent)
* Rituximab (a type of antibody)

DETAILED DESCRIPTION:
This is an open label, pilot trial of Pembrolizumab in combination with chemotherapy in participants with newly diagnosed Primary Central Nervous System Lymphoma (PCNSL).

The U.S. Food and Drug Administration (FDA) has not approved Pembrolizumab for Primary Central Nervous System Lymphoma (PCNSL) but it has been approved for other uses.

The FDA has approved Rituximab for PCNSL.

The FDA has not approved Temozolomide for PCNSL but it has been approved for other uses.

The FDA has not approved Methotrexate for PCNSL but it has been approved for other uses.

The research study procedures include screening for eligibility, blood and urine tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, testicular ultrasounds, electrocardiograms (ECG), and eye exams.

It is expected that about 15 people will take part in this research study.

Merck & Co. is supporting this research study by providing the study drug pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathologically confirmed newly diagnosed primary CNS diffuse large B-cell lymphoma (DLBCL) confirmed by one of the following:

  * Brain biopsy or resection
  * Cerebrospinal fluid
  * Vitreous fluid
* Participants must not have any evidence or history of DLBCL outside of the CNS. Participants with prior history of isolated intraocular lymphoma (primary vitreoretinal lymphoma/PVRL) who have received only local therapy are allowed.
* Participants must not have received any systemic chemotherapy or whole brain radiation therapy directed to PCNSL.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥70% will be considered if related to PCNSL, see Appendix A).
* Participants must have adequate organ function as defined below.
* Hematology

  * Absolute neutrophil count (ANC) ≥1000/µL
  * Platelets ≥100 000/µL
  * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks)
* Renal

  -- Creatinine ≤1.5 x ULN OR Measured or calculated creatinine clearance ≥40 mL/min for participant with creatinine levels >1.5 × institutional ULN (Creatinine clearance (CrCl) should be calculated per institutional standard.)
* Hepatic

  * Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 x ULN
  * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
* Coagulation

  --International normalized ratio (INR) OR prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Participants must have negative HIV serology.
* Participants must have no history of organ transplantation or ongoing immunosuppressant therapy.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative serum pregnancy within 72 hours prior to registration.
* Women in the following categories are not considered WOCBP:

  * Premenarchal
  * Premenopausal female with 1 of the following:

    * Documented hysterectomy
    * Documented bilateral salpingectomy
    * Documented bilateral oophorectomy
  * Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.
* Post-menopausal female is defined as no menses for 12 months without an alternative medical cause.

  * A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with two FSH measurements in the postmenopausal range is required.
  * Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.
* Women of child-bearing potential (WOCBP; see definition above), must agree to use a highly effective method of contraception consistently and correctly as described below during study treatment and for 120 days after study discontinuation.

  * 1. Highly Effective Contraceptive Methods That Are User Dependent (Failure rate of < 1% per year when used consistently and correctly.)

    * a. Combined (estrogen- and progestogen- containing) hormonal contraception

      * i. Oral
      * ii. Intravaginal
      * iii. Transdermal
      * iv. Injectable
    * b. Progestogen-only hormonal contraception b, c

      * i. Oral
      * ii. Injectable
  * 2. Highly Effective Methods That Have Low User Dependency (Failure rate of <1% per year when used consistently and correctly)

    * a. Progestogen- only contraceptive implant b, c
    * b. Intrauterine hormone-releasing system (IUS) b
    * c. Intrauterine device (IUD)
    * d. Bilateral tubal occlusion
    * e. Vasectomized partner: A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.
    * f. Sexual abstinence: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
* NOTES: Use should be consistent with local regulations regarding the use of contraceptive methods for participants of clinical studies.

  * a. Typical use failure rates are lower than perfect-use failure rates (i.e. when used consistently and correctly).
  * b. If hormonal contraception efficacy is potentially decreased due to interaction with study treatment, condoms must be used in addition to the hormonal contraception during the treatment period and for at least during study treatment and for 120 days after study discontinuation after the last dose of study treatment.
  * c. If locally required, in accordance with Clinical Trial Facilitation Group (CTFG) guidelines, acceptable contraceptive implants are limited to those which inhibit ovulation.
* Male participants must to use at least one of the following methods of contraception starting with the first dose of study therapy through 120 days after the last dose of therapy:

  * Be abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent
  * Use a male condom plus partner use of a contraceptive method with a failure rate of <1% per year as described in Eligibility criterion 3.1.11 when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant.
* Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile- vaginal intercourse or use a male condom during each episode of penile penetration.

Exclusion Criteria:

* Participants who cannot undergo MRI
* Intraocular PCNSL without evidence of brain or spinal cord disease.
* Participants who are receiving any other investigational agents.
* History of allergic reactions or severe hypersensitivity reactions (≥grade 3) attributed to compounds of similar chemical or biologic composition to study agent and/or any of its excipients.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137)
* Has active autoimmune disease requiring immunosuppressives or steroids
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. COVID19 vaccines are allowed.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Patient has poorly controlled diabetes mellitus with a glycosylated hemoglobin >8% or poorly controlled steroid-induced diabetes mellitus with a glycosylated hemoglobin of >8%.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction.
* Enzyme-inducing antiepileptic drugs (EIAED) need to be discontinued and switched to a non-EIAED 2 weeks prior to starting on trial drugs
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent)
* Patients who have undergone prior allogeneic stem cell transplant
* Patients who have large pleural effusions, ascites or full body edema
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Experienced Dose Limiting Toxicity (DLT) | Up to 28 days
  Dose-limiting toxicities (DLTs) will be defined as any grade ≥3 non-hematologic toxicity (with exceptions), grade 4 neutropenia lasting >7 days or febrile neutropenia, grade 4 thrombocytopenia, grade 3 thrombocytopenia with clinically significant bleeding, any grade 5 toxicity or dose delays for >14 consecutive days (related to AEs) with exceptions. Toxicities are to be assess according to the CTCAE v5.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to 16 weeks
  CRR is defined as the proportion of participants who achieved complete response (CR). Radiographic response will be assessed using IPCG criteria.
Objective Response Rate (ORR) | Up to 106 weeks
  Objective response rate (ORR), defined as best overall response of either complete or partial response, will be assessed among participants who start protocol therapy and have measurable disease at screening. Radiographic response will be assessed using IPCG criteria.
2-Year Progression Free Survival (PFS2) | Up to 2 years
  PFS2 is the percent probability estimate at 2 years based on the Kaplan-Meier method. PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy.
Duration of Response (DOR) | Up to 106 weeks
  DOR is defined as the time from date of first documented confirmed objective response to date of first documented progressive disease (PD).
Median Progression Free Survival (PFS) | Up to 106 weeks
  PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anti-cancer therapy.
Median Overall Survival (OS) | Up to 3 years
  Overall survival based on the Kaplan-Meier method is defined as the time from registration to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Frequency of Missed or Delayed doses | Up to 106 weeks
  Instances of missed or delayed doses due to treatment related toxicity will be noted to assess tolerability throughout study therapy with pembrolizumab and chemotherapy, including beyond the MTD interval.
Percentage of actual planned dosage administration | Up to 106 weeks
  Instances of actual planned cycles due to treatment related toxicity will be reported as a percentage to assess tolerability throughout study therapy with pembrolizumab and chemotherapy, including beyond the MTD interval.
Percentage of patients that discontinue study drugs due to treatment-related toxicity. | Up to 106 weeks
  Number of patients that discontinue study drugs due to treatment related toxicity; will be reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Nayak, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu